CLINICAL TRIAL: NCT02051842
Title: Effect of Metadoxine on Oxidative Stress in Non-alcoholic Fatty Liver Disease Prediabetic Mexican Patients
Brief Title: Effect of Metadoxine on Oxidative Stress in Non-alcoholic Hepatic Steatosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, Principal investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GAS-1081-13/14-1
Record Dates: First submitted 2014-01-30; First posted 2014-01-31 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: NAFLD; Pre-diabetes
Keywords: NAFLD; oxidative stress; malondialdehyde
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Glucose Intolerance | interventions — metadoxine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metadoxine (Experimental): Metadoxine 500 mg tablets by mouth every 12 hours for 6 months and metformin 500 mg tablets by mouth every 8 hours for 6 months
  Interventions: Drug: Metadoxine
- Placebo tablet (Placebo Comparator): Placebo tablet (for Metadoxine) by mouth every 12 hours for 6 months and metformin 500 mg tablets by mouth every 8 hours for 6 months
  Interventions: Drug: Metadoxine

INTERVENTIONS:
Drug: Metadoxine
  Other Names: Metadoxil; Abrixone

SUMMARY:
Oxidative stress is produced by imbalance between reactive oxygen species and antioxidant systems. This state is frequently associated with chronic diseases like obesity, insulin resistance, metabolic syndrome and hepatic steatosis. In the liver, the oxidative stress may trigger the progression of fatty liver disease, from triglyceride accumulation to inflammation, cirrhosis and hepatocellular carcinoma. Thus, the attenuation of oxidative stress, could be an important therapeutic target to lessen the severity of the disease. Until now, there is not a medical treatment to cure non-alcoholic fatty liver disease, but therapies aimed at reducing oxidative stress have been proposed. Metadoxine, an ionic complex of pyridoxine-pyrrolidone molecule, acts as a synthetic antioxidant, forming traps that can reduce free radicals; likewise, metadoxine has a proven capacity to reduce fat liver in alcoholic hepatitis. Finally, in fact that alcoholic and non-alcoholic liver diseases share molecular mechanisms in the generation of oxidative stress, the investigators propose metadoxine as a posssible modifier of the oxidative stress in non-alcoholic liver disease, prediabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* 18 to 65 years old
* Ultrasonographic diagnosis of NAFLD
* Prediabetes diagnosis

Exclusion Criteria:

* Alcoholism
* Hepatitis C or B Virus Infection
* Pregnancy
* Autoimmune hepatitis
* Metformin or metadoxine allergy
* Parenteral nutrition in the last month
* Weigh loss greater than 10% in the last month
* Taking vitamin supplements in the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress | Baseline
  Malondialdehyde levels

OTHER OUTCOMES:
Oxidative stress | 3 month follow-up
  Malondialdehyde levels
Oxidative stress | 6 months follow-up
  Malondialdehyde levels

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre, MD MSci, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán", Mexico City, Mexico